CLINICAL TRIAL: NCT03144492
Title: Microgravity Effects on Co-cultured Vascular Cells Types
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB201700297; 16-2016GL_FP-0011 (Other Grant/Funding Number: National Aeronautics and Space Administration)
Record Dates: First submitted 2017-05-02; First posted 2017-05-08 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Microgravity Exposed Endothelial Cells
Keywords: Cell Culture; Microgravity co-culture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stem cell acquisition and differentiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- self-reported healthy individuals: Self-reported healthy individuals avoiding blood draw on the days participants are feeling "under the weather"or sick. In that case, study team can delay the blood draw until the subject feels better, but this would not preclude anyone from participating.
  Interventions: Biological: Blood volume collected specifically for this study

INTERVENTIONS:
Biological: Blood volume collected specifically for this study — The subject will be sitting in a chair, and a needle will be inserted into a vein in their arm. Study Team will draw about 45ml or 3 tablespoons of whole blood for research.

SUMMARY:
The goal of this study is to assess the affect of ground based microgravity on co-cultured vascular cell types. Our goal is to better understand the cross-talk between vascular cell types grown under conditions such as microgravity as is seen in space. In this pilot study, the investigator proposes to assess changes in cell phenotype and function in microgravity as compared to normal gravity.

DETAILED DESCRIPTION:
This study builds upon previously reported space flight data in GenLab, as well as our own published data whereby the investigator evaluate the effect of microgravity on the differentiation and functional potential of circulating stem cells. The goal of this work is to leverage the powerful genetic analyses done in the SPHINX study and look at the consequences these changes have on cell-cell communications essential for vascular homeostasis, for a possible correlation to cardiovascular deconditioning. The application of this work is targeted at possible "cell based" countermeasures to address the negative effects of microgravity on the vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported healthy individuals
* Willingness to have 50mls of whole blood collected

Exclusion Criteria:

* Unwillingness to have blood used in stem cell research

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The Study team is interested in sampling a wide variety of health individuals from varying ethnic groups, sex, and age range.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Differentiation (Colony Forming) Kinetics of normal vs microgravity cultured stem cells | Within 4 weeks of collecting cells
  The study team are interesting in the effect of co-cultured Endothelial cells on the kinetics of stem cell colony formation (i.e. differentiation). As compared to normal gravity samples, the colonies that form while in co-culture with ECs will be counted and monitored. This gives a measure of the differentiation potential of these cells.

SECONDARY OUTCOMES:
Gene and Protein expression of normal vs microgravity cultured stem cells | through study completion, up to 2 years from the start of the study
  The study team will use rtPCR to probe the stem cells for the up regulation of Endothelial cell (EC) specific genes and down regulation of stem cell genes. EC specific genes include vascular endothelial cadherin (CD144), platelet endothelial cell adhesion molecule (PECAM), and von Willebrand factor (vWF). Stem cell markers include CD34. The study team will use GAPDH as a control.
Anti-thrombogenic function of normal vs microgravity cultured stem cells | through study completion, up to 2 years from the start of the study
  The study team will utilize platelet adhesion and blood clotting assays to assess any changes in how anti-thrombogenic the differentiated endothelial cells are.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Allen, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No